CLINICAL TRIAL: NCT01362738
Title: Effect of Empirical Left Atrial Appendage Isolation on Long-term Procedure Outcome in Patients With Persistent or Long-standing Persistent Atrial Fibrillation Undergoing Catheter Ablation
Acronym: BELIEF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Medical Director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCAI_BELIEF
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2016-10

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Long-standing persistent atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ablation of PV and extra-PV triggers (Active Comparator): Conventional approach which includes pulmonary vein isolation (PVI) and ablation of extra-pulmonary triggers
  Interventions: Procedure: RFCA of PV and extra-PV triggers
- LAA isolation along with the conventional ablation strategy (Active Comparator): LAA isolation along with the conventional ablation strategy
  Interventions: Procedure: LAA isolation along with the conventional ablation strategy

INTERVENTIONS:
Procedure: RFCA of PV and extra-PV triggers — PVAI and isolation of extra PV triggers
  Arms: Ablation of PV and extra-PV triggers
Procedure: LAA isolation along with the conventional ablation strategy — PVAI + isolation of extra PV triggers + LAA isolation
  Arms: LAA isolation along with the conventional ablation strategy

SUMMARY:
The purpose of this prospective randomized study is to assess whether empirical Left Atrial Appendage (LAA) isolation along with the standard approach of pulmonary vein isolation (PVI) and ablation of extra-pulmonary triggers is superior to the standard approach alone in enhancing the long-term success rate of catheter ablation in persistent or long-standing persistent atrial fibrillation (AF) patients.

DETAILED DESCRIPTION:
Persistent (PeAF) and long-standing persistent (LSP) AF are defined as sustained AFs extending beyond seven days and one year respectively (1). Hypertensive, ischemic, valvular and other structural heart diseases most commonly underlie these arrhythmias (2) and the resulting abnormal atrial substrate is believed to be the major contributor toward perpetuation of AF in these non-paroxysmal categories. Several studies have demonstrated that pulmonary vein isolation (PVI) by radiofrequency catheter ablation (RFCA) though successfully restores sinus rhythm in most patients with paroxysmal AF; it has limited success in these sustained arrhythmias (3). Presence of potential trigger-generating areas in the left and right atrium besides pulmonary veins, with reported incidence from 3.2% to 47% (4), can be held responsible for this limited success. These areas include superior vena cava, ligament of Marshall, crista terminalis, coronary sinus, left atrial (LA) posterior wall and LA appendage (3). Therefore, in order to enhance the procedural-success rate, various hybrid measures have emerged to target the PV as well as extra-PV areas that have the ability to initiate or maintain AF. Several previous studies have demonstrated the prevalence of LAA firing in patients with recurrence of AF/AT (atrial tachycardia) after catheter ablation of AF (4). Embryologically, LAA is the remnant of primitive LA, which is formed by the adsorption of primordial PV and their branches during 4th week of embryonic development. Therefore, it is logical to suggest that LAA may initiate AF like pulmonary veins. In an earlier study conducted by our group on 987 AF patients, LAA firing was revealed to be the source of AF in 27% of patients and 93% of those patients were arrhythmia free 6 months after LAA isolation (4).

Our study aims to compare the procedure outcome for two different ablation strategies; 1) standard approach of pulmonary vein isolation extended to the posterior wall down to the coronary sinus and to the left side of the interatrial septum along with isolation of superior vena cava and ablation of complex fractionated atrial electrograms (CFAE) in the atria and coronary sinus, 2) standard approach plus LAA isolation.

Hypothesis: LAA isolation combined with standard ablation procedure enhances the procedural success rate in non-paroxysmal AF patients undergoing catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years
2. History of PeAF or LSP AF refractory to antiarrhythmic drugs
3. Willing and ability to understand and sign an informed consent

Exclusion Criteria:

1. Reversible causes of AF (hyperthyroidism)
2. Left atrial thrombus
3. Moderate to severe valvular heart disease
4. Contraindication for anticoagulation
5. Life expectancy < 12 months
6. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2010-11; Primary Completion 2014-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Freedom from AF/ATs | 12 months
  Freedom from AF/ATs, defined as no episodes of AF/AT without AADs lasting >30 seconds at follow-up

SECONDARY OUTCOMES:
Severe adverse events due to cardiac cause | 12 months
  Severe adverse events (hospital admissions or death due to a cardiac cause)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation
Locations (2):
- United States (2):
  - St. David's Medical Center, Austin, Texas
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas

REFERENCES:
- [Derived] Di Biase L, Burkhardt JD, Mohanty P, Mohanty S, Sanchez JE, Trivedi C, Gunes M, Gokoglan Y, Gianni C, Horton RP, Themistoclakis S, Gallinghouse GJ, Bailey S, Zagrodzky JD, Hongo RH, Beheiry S, Santangeli P, Casella M, Dello Russo A, Al-Ahmad A, Hranitzky P, Lakkireddy D, Tondo C, Natale A. Left Atrial Appendage Isolation in Patients With Longstanding Persistent AF Undergoing Catheter Ablation: BELIEF Trial. J Am Coll Cardiol. 2016 Nov 1;68(18):1929-1940. doi: 10.1016/j.jacc.2016.07.770. PMID 27788847